CLINICAL TRIAL: NCT06537050
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of JX2105 in Healthy Chinese Subjects The Purpose of the Study is to Evaluate the Safety, Tolerability After Administration of Single Dose or Multiple Doses, and the Pharmacokinetics (PK) of Single and Multiple Doses of JX2105 in Healthy Study Participants.
Brief Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of JX2105 in Healthy Chinese Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Jingxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JX2105-I-01
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JX2105 (Active Comparator): JX2105 10mg；JX2105 30mg；JX2105 90mg；JX2105 180mg
  Interventions: Drug: JX2105
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JX2105 — Oral capsule
  Arms: JX2105
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability after administration of single dose or multiple doses, and the pharmacokinetics (PK) of single and multiple doses of JX2105 in healthy study participants.

DETAILED DESCRIPTION:
Overall design:

This study is divided into 3 parts: Part 1: single-dose escalation study (SAD); Part 2: multiple-dose escalation study (MAD); Part 3: food-effect study (FE). Part 1 includes 7 cohorts; Part 2 includes 2~3cohorts; and Part 3 food effect study will conduct on 1 dose strength to evaluate the effect of food intake on pharmacokinetic/pharmacodynamics of JX2105 and its metabolites. The doses of part 2 and 3 will be designed according to the PK parameters from Part 1. Maximum recommended human dose of part 1 is 10 mg and the maximum dose is 180 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy participant must be 18 to 75 years of age inclusive.
2. Body mass index (BMI) within the range 18.5 to 28 kg/m^2 (inclusive).
3. Subjects must adhere to contraception restrictions from signing the informed consent to 3 months after the last dose.
4. Willing to participate in the clinical trial and provide signed informed consent.

Exclusion Criteria:

1. Having a history or present condition of diseases or dysfunction that may affect the clinical trial on the consideration of investigator, including but not limited to central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, blood system and other diseases;
2. Having a history or present condition of mental illness;
3. Any surgical condition or condition that could significantly affect the absorption, distribution, metabolism, and excretion of the investigational drug or could jeopardize the subjects participating in the trial; such as a history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcer, gastrointestinal bleeding, etc.;
4. Usage of any drugs within 2 weeks before screening, including prescription drugs, over-the-counter drugs and Chinese herbal medicines;
5. With a known history of allergy to investigational drug ingredients or similar drugs, history of allergic diseases or allergic constitution;
6. Having clinical significance in laboratory test in the opinion of the Investigator, or creatinine clearance < 80 mL/min;
7. Having clinical significant electrocardiogram (ECG) abnormality and chest X-ray examination indicators, in the opinion of the Investigator;
8. Having clinical significance in vital signs, with sitting resting pulse rate < 50 beats/min or > 100 beats/min; systolic blood pressure < 90 mmHg or > 140 mmHg; diastolic blood pressure < 50 mmHg or > 90 mmHg, in the opinion of the Investigator;
9. Having one or more clinically significant tests for hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antibody and treponema pallidum antibody;
10. Female participant with positive pregnancy test results;
11. History of drug or drug abuse within 1 year before screening, or positive urine drug screening;
12. Alcohol abuse within 1 year before screening, with an average weekly alcohol intake of more than 14 units or positive alcohol breath test;
13. With average daily smoking ≥ 5 cigarettes within 3 months before screening;
14. With no suitable veins for multiple venipuncture/catheterization as assessed at screening;
15. Having blood donation (including blood component donation) or massive blood loss (≥ 200 mL) within 3 months before screening; or receive blood transfusion or using blood products;
16. Having a history of surgery within 3 months before screening, or has not recovered from surgery, or will have a scheduled surgery during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
TEAE/SAE | Day1 to Day 10
  The number, frequency and incidence of TEAE/SAE; The number, frequency and incidence of drug-related TEAE/SAE;

SECONDARY OUTCOMES:
Cmax | Day1 to Day 10
  Peak concentrations (Cmax) of JX2105 and metabolites detected after administration; Area under the drug concentration-time curve (AUC0-last) from 0h to the last sample collection time t where the concentration of JX2105 and metabolites can be accurately determined;
AUC0-∞ | Day1 to Day 10
  Area under the drug concentration-time curve of JX2105 and metabolites from 0 to infinity (AUC0-∞)
Tmax | Day1 to Day 10
  Peak time of JX2105 and its metabolites
t1/2z | Day1 to Day 10
  End phase elimination half-life
λz | Day1 to Day 10
  End-phase elimination rate constant
Vz/F | Day1 to Day 10
  Apparent volume of distribution
CLz/F | Day1 to Day 10
  Apparent clearance
MRT0-last、 MRT0-∞ | Day1 to Day 10
  Mean residence time

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China